CLINICAL TRIAL: NCT02284178
Title: Oral Suction Intervention to Reduce Aspiration and Ventilator Events: NO-ASPIRATE
Acronym: NO-ASPIRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Orlando Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R01NR014508-01A1 (NIH)
Record Dates: First submitted 2014-10-15; First posted 2014-11-05 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; aspiration; suctioning; secretions; ventilator-associated events
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced oral suction (Experimental): Deep oropharyngeal suction with catheter
  Interventions: Other: Enhanced oropharyngeal suction
- Usual Care Oral Suction (Sham Comparator): Oropharyngeal suction with suction swab
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Enhanced oropharyngeal suction — Deep oropharyngeal suction with catheter every 4 hours
  Arms: Enhanced oral suction
Other: Usual Care — Oral suction with suction swab every 4 hours
  Arms: Usual Care Oral Suction

SUMMARY:
Insertion of a breathing tube to enable treatment with mechanical ventilation (respirator) is often associated with complications, such as infection and lung injury. Leakage of secretions around the breathing tube (microaspiration) is a major factor leading to complications. The investigators propose that a standardized, enhanced oral suction protocol will be effective in reducing microaspiration and harms associated with mechanical ventilation. The investigators hypothesize that those randomized to the enhanced oral suction protocol will have less microaspiration and other ventilator-associated conditions than those in the usual care, standard suction group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* orally intubated with endotracheal tube and treated with mechanical ventilation
* 24 hours or less since intubation
* expected to be intubated for at least 36 hours after enrollment

Exclusion Criteria:

* documented aspiration at time of intubation
* intubation to treat known aspiration
* treatment with rescue mechanical ventilation therapies (oscillator)
* re-intubation
* contraindications to receiving the intervention (e.g., oral injuries)
* history of lung or head/neck cancers that may produce amylase in the lungs
* history of disease that affects saliva production (e.g., Sjögren's syndrome)
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Sole, PhD, Principal Investigator — Univesity of Central Florida
Locations (1):
- Orlando Regional Medical Center, Orlando, Florida, United States

REFERENCES:
- [Derived] Bourgault AM, Xie R, Talbert S, Sole ML. Association of enteral feeding with microaspiration in critically ill adults. Appl Nurs Res. 2022 Oct;67:151611. doi: 10.1016/j.apnr.2022.151611. Epub 2022 Jun 30. PMID 36116866
- [Derived] Talbert S, Bourgault AM, Rathbun KP, Abomoelak B, Deb C, Mehta D, Sole ML. Pepsin A in Tracheal Secretions From Patients Receiving Mechanical Ventilation. Am J Crit Care. 2021 Nov 1;30(6):443-450. doi: 10.4037/ajcc2021528. PMID 34719715
- [Derived] Sole ML, Talbert S, Yan X, Penoyer D, Mehta D, Bennett M, Emery KP, Middleton A, Deaton L, Abomoelak B, Deb C. Impact of deep oropharyngeal suctioning on microaspiration, ventilator events, and clinical outcomes: A randomized clinical trial. J Adv Nurs. 2019 Nov;75(11):3045-3057. doi: 10.1111/jan.14142. Epub 2019 Aug 7. PMID 31241194

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Oral Suction: Deep oropharyngeal suction with catheter every 4 hours; standard oral cleansing every 4 hours.
- Usual Care Oral Suction: Oral suction with suction swab every 4 hours; standard oral cleansing every 4 hours.
Period: Overall Study
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Started | 255 | 258
Completed | 206 | 204
Not Completed | 49 | 54
Not completed — Met exclusion criteria | 49 | 54

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Oral Suction: Oropharyngeal suction with suction swab; standard oral cleansing every 4 hours.
- Total: Total of all reporting groups
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction | Total
Number analyzed (Participants) | 255 | 258 | 513
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.05 (18.93) | 57.50 (18.69) | 58.77 (18.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 112 | 217
  Male | 150 | 146 | 296
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 43 | 95
  Not Hispanic or Latino | 203 | 215 | 418
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 15 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 54 | 104
  White | 196 | 186 | 382
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 255 | 258 | 513
APACHE 2 [Mean (Standard Deviation); unit: units on a scale] — Severity of illness; Range 0-71; higher number = greater severity; rare for scores to exceed 55
  units on a scale | 22.98 (7.21) | 22.72 (7.94) | 22.85 (7.58)

OUTCOME MEASURES:

1. Primary Outcome: Microaspiration as Measured by Tracheal Amylase
Description: Specimens will be obtained every 12 hours for up to 14 days or subject no longer meets inclusion (e.g., extubation, tracheostomy, etc.); tracheal amylase measured in U/L.
Time Frame: Every 12 hours up to 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
U/L | 13,086 (25,288) | 15,298 (36,643)
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.432, GEE analysis

2. Primary Outcome: Microaspiration as Measured by Percentage of Tracheal Specimens Positive for Amylase Per Participant
Description: Specimens will be obtained every 12 hours for up to 14 days or subject no longer meets inclusion criteria
Time Frame: Every 12 hours up to 14 days
Measure: Number; unit: percentage specimens positive amylase
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
percentage specimens positive amylase | 75.2 | 78.4
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.684, GEE

3. Secondary Outcome: Ventilator-Associated Condition (VAC) Rate
Description: VAC rate was calculated between control and intervention groups using the Centers for Disease Control and Prevention (2013) criteria.
Time Frame: VAC assessed for 2 days beyond last intervention; mean 5.4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
Participants | 31 | 32
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.858, Chi-squared

4. Secondary Outcome: Time to VAC
Time Frame: VAC was assessed for two days beyond the last intervention; mean 5.4 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
Days | 4.94 (2.29) | 5.72 (2.53)

5. Other Pre Specified Outcome: Tracheal to Oral Ratio of Amylase
Description: The ratio of the tracheal value to the oral value of amylase for each paired sample was calculated (ratio included baseline specimen collected).
Time Frame: Every 12 hours up to 14 days
Measure: Mean (Standard Deviation); unit: Ratio of tracheal amylase to oral value
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
Ratio of tracheal amylase to oral value | 0.073 (0.1) | 0.075 (0.2)
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.460, GEE analysis

6. Post Hoc Outcome: Clinical Outcome: Ventilator Hours
Time Frame: Duration of Mechanical Ventilation
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
Hours | 147.6 (86.4) | 159.3 (102.6)
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.214, t-test, 2 sided

7. Post Hoc Outcome: Clinical Outcome: Intensive Care Unit Length of Stay
Time Frame: Duration of Intensive Care Unit Stay
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
Days | 9.8 (6.6) | 10.8 (7.7)
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.155, t-test, 2 sided

8. Post Hoc Outcome: Clinical Outcome: Hospital Length of Stay
Time Frame: Duration of Hospital Stay
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
Number analyzed (Participants) | 206 | 204
Days | 19.5 (16.5) | 23.4 (23.1)
Statistical Analysis 1: Comparison: Enhanced Oral Suction vs Usual Care Oral Suction; Test type: Superiority; p = 0.050, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Data were collected for the duration of participant enrollment in study (mean 5.4 days); range 1.5 to 14.0 days.
Arm/Group | Enhanced Oral Suction | Usual Care Oral Suction
All-Cause Mortality (participants affected / at risk) | 41/206 | 49/204
Serious Adverse Events (participants affected / at risk) | 0/206 | 0/204
Other Adverse Events (participants affected / at risk) | 0/206 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT02284178/Prot_SAP_000.pdf